CLINICAL TRIAL: NCT03686371
Title: Evaluation of Pain Following Scoliosis Surgery.- RACHIDOL
Brief Title: Evaluation of Pain Following Scoliosis Surgery.
Acronym: RACHIDOL
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC17_3088_RACHIDOL
Record Dates: First submitted 2018-09-10; First posted 2018-09-26 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Idiopathic Scoliosis
MeSH Terms: interventions — Spinal Fusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: posterior surgery for spinal arthrodesis — posterior surgery for spinal arthrodesis

SUMMARY:
The main objective of this study was to evaluate acute pain following scoliosis surgery in adolescent.

ELIGIBILITY:
Inclusion Criteria:

* adolescent from 10 to 18 years of age
* idiopathic scoliosis
* posterior surgery for spinal arthrodesis
* non opposition children and parents

Exclusion Criteria:

* complication following surgery needing reoperation
* secondary intervention
* anterior surgery
* non idiopathic scoliosis

Ages: 10 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: adolescent with scoliosis surgery for idiopathic scoliosis
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-10-23 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Visual Analog Score for pain (EVA) | 3 days after inclusion
  The assessment criteria used is the numerical pain scale from 0 to 10(0 = no pain, 10 = extremely painful

CONTACTS AND LOCATIONS:
Overall Officials: Anne DEFONTAINE, MD, Principal Investigator — Rennes University Hospital
Locations (1):
- CHU de Rennes, Rennes, France